CLINICAL TRIAL: NCT04567680
Title: Acceptance and Commitment Therapy to Improve Social Support for Veterans With PTSD
Acronym: ACT-SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3382-R; 1I01RX003382-01A1 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; Social Support; Veterans; Social Functioning; Community Reintegration
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Social Adjustment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent evaluator will assess outcomes for each study participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and Commitment Therapy to Improve Social Support (Experimental): This treatment is designed to help Veterans with PTSD increase social support in family, partner, and peer relationships by reducing experiential avoidance. ACT-SS is specifically designed to address deficits in the entire social support network for Veterans with PTSD.
  Interventions: Behavioral: Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD
- Present-Centered Therapy (Active Comparator): PCT is designed to provide the emotional support for individuals with PTSD that will assist with recovery. The focus of PCT is on the "here and now," including current life difficulties that are directly or indirectly related to the experience of trauma. PCT aims to help the patient consider ways to react to these difficulties.
  Interventions: Behavioral: Present-Centered Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD — This treatment is designed to help Veterans with PTSD increase social support in family, partner, and peer relationships by reducing experiential avoidance. ACT-SS is specifically designed to address deficits in the entire social support network for Veterans with PTSD.
  Other Names: ACT-SS
  Arms: Acceptance and Commitment Therapy to Improve Social Support
Behavioral: Present-Centered Therapy — PCT is designed to provide the emotional support for individuals with PTSD that will assist with recovery. The focus of PCT is on the "here and now," including current life difficulties that are directly or indirectly related to the experience of trauma. PCT aims to help the patient consider ways to react to these difficulties.
  Other Names: PCT
  Arms: Present-Centered Therapy

SUMMARY:
Veterans with PTSD often have impaired social relationships and poor social support. The negative outcomes associated with poor social support are of particular concern for Veterans with PTSD, who often perceive the world to be dangerous, view their social support network as a threat to their safety, and avoid members of their support network in order to increase their perceived safety. The goal of this project is to evaluate the efficacy of Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD (ACT-SS), a treatment focused on helping Veterans with PTSD to increase social support with family relationships, partners, and peers by targeting maladaptive patterns of interpersonal difficulties, feelings of detachment from others, irritability, and avoidance of social situations. The primary aim of this study is to conduct a two-site randomized controlled trial of ACT-SS (n=75) vs. PCT (n=75), a common treatment for social support difficulties. If positive, this study will provide a critically-needed treatment for Veterans with PTSD to improve their social functioning and social reintegration in the community.

DETAILED DESCRIPTION:
Veterans with PTSD often have substantial interpersonal problems and low perceived social support from family, partners, and peers. Interpersonal problems result in poor social reintegration, which in turn permeates all aspects of their functioning and is associated with greater suicidal ideation. The problems emerge rapidly, with one study showing a fourfold increase in rates of self-reported interpersonal conflict within six months of returning from deployment. Veterans with PTSD report considerable avoidance in relationships, marital stress, intimacy difficulties, and parenting problems. Low social support is a key factor related to poor physical health, emotional functioning, and increased mortality risk. Given the importance of social relationships in buffering against negative outcomes and suicidal ideation for persons with PTSD, there is a strong need for more research and treatment development to improve the social functioning of these Veterans. The proposed project will focus on evaluating an innovative treatment for improving the social relationships and social support among Veterans with PTSD.

The goal of this project is to evaluate the efficacy of Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD (ACT-SS), a treatment focused on helping Veterans with PTSD to increase social support with family relationships, partners, and peers by targeting maladaptive patterns of interpersonal difficulties, feelings of detachment from others, irritability, and avoidance of social situations. ACT-SS provides Veterans with PTSD with more adaptive coping skills (i.e., acceptance and mindfulness, focus on values-based living) to improve social relationships, social support, and help manage PTSD-related distress. The investigators' pilot data of ACT-SS indicates that ACT-SS results in improved social relationships and reduced PTSD symptoms, with preliminary data showing that ACT-SS results in significantly better improvement in social functioning outcomes compared to Present-Centered Therapy (PCT).

The primary aim of this study is to conduct a two-site randomized controlled trial of ACT-SS (n=75) vs. PCT (n=75), a common treatment for social support difficulties. Study outcomes will include measures of social support, social relationships, quality of life, and PTSD symptoms. This proposal, supported by the promising pilot data, represents an important step in examining the potential efficacy of ACT-SS, including social functioning and quality of life in Veterans with PTSD. If positive, results from this study may provide a new treatment approach for improving the social reintegration of Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-5 PTSD diagnosis
* Minimum score of 31 on the PCL-5
* Clinically significant difficulties in interpersonal relationships
* Competent to provide written informed consent
* Ages 18 and older
* If being treated with psychoactive medication, no change in drugs or dose for the past 2 months
* Willingness to be audio-taped

Exclusion Criteria:

* Any current or lifetime DSM-5 psychotic disorder
* Current or recent (within 1 month of study entry) DSM-5 substance use disorder
* Cognitive impairment that would interfere with study participation
* Current manic episode
* Recent clinically significant suicidality (past 3 months)
* Moderate to severe domestic violence (measured by the Conflict Tactics Scale-2)
* Current PTSD psychotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in the Social Adjustment Scale-Self Report | Baseline, End of Treatment (12 weeks), 3-month follow-up, and 6-month follow-up
  The Social Adjustment Scale-Self Report (SAS-SR) is a 54-item measure of current social functioning in 6 domains: Work; Social and Leisure; Extended Family; Primary Relationship; Parental; and Family Unit. It is the primary measure of change in social functioning for the study. An Overall Adjustment scale provides a total score (alpha = .74-.85; test-retest r's = .78-.80). The SAS-SR is sensitive to change and has good convergent and discriminant validity. Higher scores indicate better functioning. Scores for each role area are calculated by averaging the scores for all answered items within that area. The total score is calculated by averaging all applicable items.
Change in the MOS Social Support Survey | Baseline, End of Treatment (12 weeks), 3-month follow-up, and 6-month follow-up
  Social Support: The MOS Social Support Survey is a 19-item multidimensional, self-administered survey of social support for individuals with chronic conditions. It includes four functional support scales, including emotional/informational, tangible, affectionate, and positive social interaction. Scores range from 0-100. A higher score for an individual scale or for the overall support index indicates more support.

SECONDARY OUTCOMES:
Change in the Quality of Life, Enjoyment, and Satisfaction Questionnaire | Baseline, End of Treatment (12 weeks), 3-month follow-up, and 6-month follow-up
  Quality of Life: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a commonly used self-report measure to assess quality of life in several domains: general activities, physical health, subjective feelings, leisure time activities, social relationships, work, and household duties. The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70. Percent maximum scores range from 0-100. Higher scores indicating greater life satisfaction and enjoyment.
Change in the Clinician Administered PTSD Scale (CAPS-5) | Baseline, End of Treatment (12 weeks), 3-month follow-up, and 6-month follow-up
  The Clinician Administered PTSD Scale (CAPS-5) is a structured interview that will be used to diagnose PTSD and to obtain data (pre and post treatment, follow-up) on the frequency and severity of PTSD symptoms. The CAPS-5 is the gold standard for assessing PTSD. CAPS-5 scores range from 0 to 80 with higher scores indicating greater PTSD symptom severity.
Change in the PTSD Checklist (PCL-5) | Baseline, End of Treatment (12 weeks), 3-month follow-up, and 6-month follow-up
  The PCL-5 is a 20-item self-report measure of PTSD symptoms, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Marie Kelly, PhD MS, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Final data sets from the study, composed of de-identified data, will be archived and available to others by request to the PI. All publications from this study will be made available to the public through the National Library of Medicine PubMed Central website within one year after the research article is published.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the project has ended and will be available for seven years after the project has closed.

DOCUMENTS (1):
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT04567680/ICF_000.pdf